CLINICAL TRIAL: NCT00471276
Title: A Phase II Study Of Sunitinib Malate Single Agent For The Treatment Of Women With Advanced Breast Cancer
Brief Title: Efficacy And Safety Of Sunitinib In Women With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181068
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Results first posted 2011-07-22 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Breast Neoplasms
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — sunitinib (Sutent), 37.5 mg, daily dosing
  Other Names: Sutent, sunitinib

SUMMARY:
Patients with advanced breast cancer to receive sunitinib (Sutent) once daily until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of breast cancer
* Metastatic or locally recurrent disease that is, in the opinion of the investigator, not amenable to resection or radiation therapy
* Patients with at least one measurable lesion as per RECIST

Exclusion Criteria:

* Inflammatory breast cancer
* Prior treatment with VEGF inhibitors (unless in adjuvant setting at least 12 months ago)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- United States (27):
  - Pfizer Investigational Site, Bakersfield, California
  - Pfizer Investigational Site, Burbank, California
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Hawthorne, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Boynton Beach, Florida
  - Pfizer Investigational Site, Zion, Illinois
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Maple Grove, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Kernersville, North Carolina
  - Pfizer Investigational Site, Lexington, North Carolina
  - Pfizer Investigational Site, North Wilkesboro, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Smyrna, Tennessee
  - Pfizer Investigational Site, Everett, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181068&StudyName=Efficacy%20And%20Safety%20Of%20Sunitinib%20In%20Women%20With%20Advanced%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: Sunitinib 37.5 milligrams (mg) daily by oral capsule in continuous daily dose (CDD) schedule. Dose adjustments, if needed, included a reduction to 25mg daily or escalation to 50mg daily anytime after Week 12.
Period: Overall Study
Arm/Group | Sunitinib
Started | 83
Completed | 0
Not Completed | 83
Not completed — Death | 2
Not completed — Adverse Event | 16
Not completed — Protocol Violation | 1
Not completed — Objective progression or relapse | 54
Not completed — Global deterioration of health status | 1
Not completed — Other | 3
Not completed — Refused treatment | 6

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 83
Age Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Number of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR defined as disappearance of all target lesions. PR defined as a greater than or equal to 30 percent (≥30%) decrease in sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline, Week 9, and every 8 weeks up to Month 34
Population: Intent to Treat (ITT) population: all enrolled participants
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 83
Participants | 7
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; Exact 2-sided confidence interval; Objective Response Rate (percent) = 8.4, 95% CI 2-sided [3.5 to 16.6]

2. Secondary Outcome: Number of Participants With Clinical Benefit
Description: The sum of participants with confirmed CR, PR, and stable disease (SD) greater than (>) 6 months according to RECIST. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference smallest sum of longest dimensions since treatment started.
Time Frame: Baseline, Week 9, and every 8 weeks up to Month 34
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 83
Participants | 9
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; Exact 2-sided confidence interval; Objective Response Rate (percent) = 10.8, 95% CI 2-sided [5.1 to 19.6]

3. Secondary Outcome: Number of Participants With Objective Response of Superficial Lesions
Description: Number of participants with objective response based assessment of confirmed CR or PR of superficial lesions according to RECIST. Superficial lesions included skin lesions, chest wall lesions, and breast lesions and lymph nodes if followed up by physical examination.
Time Frame: Baseline, every 4 weeks up to Month 34
Population: ITT; Number of participants analyzed equaled (N =) participants who had superficial lesions with post baseline follow-up assessments of those lesions.
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 15
Participants | 3

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time from date of randomization to date of first documentation of objective tumor progression or death due to any cause, whichever occurred first. PFS calculated as (Months)=(first event date minus randomization date plus 1) divided by 30.4.
Time Frame: Baseline up to Month 34
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 83
Months | 3.6 [2.4 to 3.9]

5. Secondary Outcome: Duration of Response (DR)
Description: Time from first objective documentation of complete or partial response that was subsequently confirmed to first documentation of disease progression or death due to any cause, whichever occurred first. DR calculated as (Weeks)=(end date for DR minus first subsequent confirmed CR or PR plus 1) divided by 7.
Time Frame: Baseline up to Month 34 or early termination
Population: ITT; N=participants with objective response
Measure: Median (Full Range); unit: Weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 7
Weeks | 3.4 [1.9 to 12.9]

6. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to date of death due to any cause. OS (Months)=(death date minus date of first dose of study medication plus 1) divided by 30.4. For participants who were alive, overall survival was censored at last contact.
Time Frame: Baseline until death (up to Month 34)
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 83
Months | 15.6 [14.0 to 22.7]

7. Secondary Outcome: Number of Participants With Objective Response for Subgroup of Participants Whom Sunitinib Was at Least a Third Line Therapy
Description: Number of participants with objective response based assessment of confirmed CR or PR according to RECIST. CR defined as disappearance of all target lesions. PR defined as ≥30% decrease in sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline, Week 9, and every 8 weeks up to Month 34
Population: ITT; N=participants who received at least 2 lines of prior chemotherapy for advanced/metastatic disease and had post baseline tumor assessment
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 3
Participants | 1

8. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionaire-C30 (EORTC- QLQ-C30) Score
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms. Change from baseline=Cycle/Day score minus baseline score.
Time Frame: Baseline, every 4 weeks up to Month 31 or early termination
Population: ITT; N=participants who completed the scales at both baseline and any cycle; n=number of participants who completed the scales at both baseline and the respective cycle. Results reported for Cycles 1 through 6 only, because (n) decreased substantially after Cycle 6.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 76
Units on a scale
  Week 4 (Cycle 2/Day 1) (n=64) | 0.0 [-83 to 100]
  Month 2 (Cycle 3/Day 1) (n=44) | -8.3 [-67 to 75]
  Month 3 (Cycle 4/Day 1) (n=34) | -16.7 [-75 to 66.7]
  Month 4 (Cycle 5/Day 1) (n=19) | -8.3 [-67 to 66.7]
  Month 5 (Cycle 6/Day 1) (n=16) | -8.3 [-42 to 33.3]
  Baseline (Cycle 1/Day 1) (n=76) | 66.7 [0 to 100]

9. Secondary Outcome: Change From Baseline in EORTC-QLQ Companion Breast Cancer Module (EORTC-QLQ-BR23) Score: Body Image
Description: EORTC-QLQ-BR23: included functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and single item symptoms scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). Questions used 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Scores averaged and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems. Change from baseline=Cycle/Day score minus baseline score.
Time Frame: Baseline, every 4 weeks up to Month 31 or early termination
Population: as for outcome 8
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 77
Units on a scale
  Week 4 (Cycle 2/Day 1) (n=60) | 0.0 [-42 to 66.7]
  Month 2 (Cycle 3/Day 1) (n=38) | 0.0 [-33 to 91.7]
  Month 3 (Cycle 4/Day 1) (n=29) | 0.0 [-75 to 91.7]
  Month 4 (Cycle 5/Day 1) (n=17) | 0.0 [-33 to 16.7]
  Month 5 (Cycle 6/Day 1) (n=14) | 0.0 [-42 to 8.33]
  Baseline (Cycle 1/Day 1) (n=77) | 83.3 [0 to 100]

10. Secondary Outcome: Change From Baseline in EORTC-QLQ-BR23 Score: Future Perspective
Description: as for outcome 9
Time Frame: Baseline, every 4 weeks up to Month 31 or early termination
Population: as for outcome 8
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 76
Units on a scale
  Week 4 (Cycle 2/Day 1) (n=59) | 0.0 [-100 to 66.7]
  Month 2 (Cycle 3/Day 1) (n=38) | -33.3 [-100 to 33.3]
  Month 3 (Cycle 4/Day 1) (n=29) | -33.3 [-100 to 33.3]
  Month 4 (Cycle 5/Day 1) (n=17) | 0.0 [-67 to 0]
  Month 5 (Cycle 6/Day 1) (n=14) | -16.7 [-67 to 33.3]
  Baseline (Cycle 1/Day 1) (n=76) | 66.7 [0 to 100]

11. Secondary Outcome: Change From Baseline in EORTC-QLQ-BR23 Score: Sexual Enjoyment
Description: as for outcome 9
Time Frame: Baseline, every 4 weeks up to Month 31 or early termination
Population: as for outcome 8
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 32
Units on a scale
  Week 4 (Cycle 2/Day 1) (n=17) | 0.0 [-33 to 100]
  Month 2 (Cycle 3/Day 1) (n=10) | 0.0 [-33 to 33.3]
  Month 3 (Cycle 4/Day 1) (n=6) | 0.0 [-67 to 33.3]
  Month 4 (Cycle 5/Day 1) (n=5) | 0.0 [0 to 66.7]
  Month 5 (Cycle 6/Day 1) (n=4) | 0.0 [0 to 100]
  Baseline (Cycle 1/Day 1) (n=32) | 33.3 [0 to 100]

12. Secondary Outcome: Change From Baseline in EORTC-QLQ-BR23 Score: Sexual Functioning
Description: as for outcome 9
Time Frame: Baseline, every 4 weeks up to Month 31 or early termination
Population: as for outcome 8
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 72
Units on a scale
  Week 4 (Cycle 2/Day 1) (n=56) | 0.0 [-33 to 100]
  Month 2 (Cycle 3/Day 1) (n=36) | 0.0 [-83 to 33.3]
  Month 3 (Cycle 4/Day 1) (n=25) | 0.0 [-100 to 16.7]
  Month 4 (Cycle 5/Day 1) (n=15) | 0.0 [-33 to 0]
  Month 5 (Cycle 6/Day 1) (n=12) | 0.0 [-33 to 0]
  Baseline (Cycle 1/Day 1) (n=72) | 100.0 [0 to 100]

13. Secondary Outcome: Change From Baseline in EORTC-QLQ-BR23 Score: Arm Symptoms
Description: as for outcome 9
Time Frame: Baseline, every 4 weeks up to Month 31 or early termination
Population: as for outcome 8
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 77
Units on a scale
  Week 4 (Cycle 2/Day 1) (n=62) | 0.0 [-67 to 44.4]
  Month 2 (Cycle 3/Day 1) (n=40) | 0.0 [-67 to 44.4]
  Month 3 (Cycle 4/Day 1) (n=30) | 0.0 [-67 to 44.4]
  Month 4 (Cycle 5/Day 1) (n=17) | 0.0 [-67 to 66.7]
  Month 5 (Cycle 6/Day 1) (n=14) | 0.0 [-67 to 33.3]
  Baseline (Cycle 1/Day 1) (n=77) | 11.1 [0 to 77.8]

14. Secondary Outcome: Change From Baseline in EORTC-QLQ-BR23 Score: Breast Symptoms
Description: as for outcome 9
Time Frame: Baseline, every 4 weeks up to Month 31 or early termination
Population: as for outcome 8
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 76
Units on a scale
  Week 4 (Cycle 2/Day 1) (n=61) | 0.0 [-42 to 33.3]
  Month 2 (Cycle 3/Day 1) (n=39) | 0.0 [-42 to 16.7]
  Month 3 (Cycle 4/Day 1) (n=30) | 0.0 [-50 to 33.3]
  Month 4 (Cycle 5/Day 1) (n=17) | 0.0 [-50 to 13.9]
  Month 5 (Cycle 6/Day 1) (n=14) | 0.0 [-42 to 8.33]
  Baseline (Cycle 1/Day 1) (n=76) | 8.3 [0 to 83.3]

15. Secondary Outcome: Change From Baseline in EORTC-QLQ-BR23 Score: Systemic Therapy Side Effects
Description: as for outcome 9
Time Frame: Baseline, every 4 weeks up to Month 31 or early termination
Population: as for outcome 8
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 77
Units on a scale
  Week 4 (Cycle 2/Day 1) (n=62) | 14.3 [-24 to 57.1]
  Month 2 (Cycle 3/Day 1) (n=40) | 19.0 [-24 to 52.4]
  Month 3 (Cycle 4/Day 1) (n=29) | 14.3 [-14 to 57.1]
  Month 4 (Cycle 5/Day 1) (n=17) | 23.8 [-4.8 to 61.9]
  Month 5 (Cycle 6/Day 1) (n=14) | 19.0 [4.76 to 42.9]
  Baseline (Cycle 1/Day 1) (n=77) | 14.3 [0 to 76.2]

16. Secondary Outcome: Change From Baseline in EORTC-QLQ-BR23 Score: Upset by Hair Loss
Description: as for outcome 9
Time Frame: Baseline, every 4 weeks up to Month 31 or early termination
Population: as for outcome 8
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 25
Units on a scale
  Week 4 (Cycle 2/Day 1) (n=5) | 0.0 [-33 to 33.3]
  Month 2 (Cycle 3/Day 1) (n=8) | 0.0 [0 to 0]
  Month 3 (Cycle 4/Day 1) (n=6) | 0.0 [0 to 100]
  Month 4 (Cycle 5/Day 1) (n=5) | 0.0 [0 to 100]
  Month 5 (Cycle 6/Day 1) (n=4) | 0.0 [0 to 66.7]
  Baseline (Cycle 1/Day 1) (n=25) | 0.0 [0 to 100]

17. Secondary Outcome: Change From Baseline in Cancer Therapy Satisfaction Questionnaire (CTSQ) Score: Expectation of Therapy
Description: CTSQ: included 3 multi-item subscales (Expectation of Therapy [ET], Satisfaction with Therapy [SWT], and Feelings about Side Effects [FSE]). Questions used 5-point scale from 1 'Never' to 5 'Always'. Scores averaged and transformed to 0-100 scale, with higher scores associated with better outcomes. Change from baseline=score for Cycle/Day minus baseline score.
Time Frame: Baseline, Day 15, Week 4 and 8, and every 8 weeks up to Month 36 or early termination
Population: ITT; N=participants with baseline CTSQ data and data on any cycle/day; n=participants with baseline CTSQ data and data at corresponding cycle/day. Cycle 1 Day 15 measurements only for subset of participants with loco-regional superficial disease. Results reported for Cycles 1, 2, 3, 5 and 7 only, because (n) decreased substantially after Cycle 7.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 59
Units on a scale
  Baseline (Cycle 1/Day 1) (n=59) | 70.00 [0.00 to 100.0]
  Cycle 1/Day 15 (n=2) | 20.00 [10.00 to 30.00]
  Week 4 (Cycle 2/Day 1) (n=48) | 0.00 [-35.0 to 75.00]
  Week 8 (Cycle 3/Day 1) (n=31) | 5.00 [-50.0 to 75.00]
  Month 4 (Cycle 5/Day 1) (n=11) | 5.00 [-30.0 to 35.00]
  Month 6 (Cycle 7/Day 1) (n=2) | 17.50 [0.00 to 35.00]

18. Secondary Outcome: Change From Baseline in CTSQ Score: Feelings About Side Effects
Description: as for outcome 17
Time Frame: Baseline, Day 15, Week 4 and 8, and every 8 weeks up to Month 36 or early termination
Population: as for outcome 17
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 58
Units on a scale
  Cycle 1/Day 15 (n=2) | 3.13 [-12.5 to 18.75]
  Week 4 (Cycle 2/Day 1) (n=47) | 0.00 [-56.3 to 75.00]
  Week 8 (Cycle 3/Day 1) (n=31) | 0.00 [-62.5 to 75.00]
  Month 4 (Cycle 5/Day 1) (n=12) | 0.00 [-56.3 to 75.00]
  Month 6 (Cycle 7/Day 1) (n=2) | -6.25 [-18.8 to 6.25]
  Baseline (Cycle 1/Day 1) (n=58) | 62.50 [12.50 to 100.0]

19. Secondary Outcome: Change From Baseline in CTSQ Score: Satisfaction With Therapy
Description: as for outcome 17
Time Frame: Baseline, Day 15, Week 4 and 8, and every 8 weeks up to Month 36 or early termination
Population: as for outcome 17
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 59
Units on a scale
  Cycle 1/Day 15 (n=2) | 8.93 [0.00 to 17.86]
  Week 4 (Cycle 2/Day 1) (n=48) | 10.71 [-35.7 to 53.57]
  Week 8 (Cycle 3/Day 1) (n=31) | 7.14 [-58.9 to 60.71]
  Month 4 (Cycle 5/Day 1) (n=12) | 11.79 [-32.1 to 57.14]
  Month 6 (Cycle 7/Day 1) (n=2) | -1.79 [-3.57 to 0.00]
  Baseline (Cycle 1/Day 1) (n=59) | 71.43 [25.00 to 100.0]

20. Other Pre Specified Outcome: 1-Year Survival Probability
Description: Probability of survival 1 year after the first dose of study treatment.
Time Frame: Baseline up to 1 year
Population: ITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 83
Percentage of participants | 65.0 [54.5 to 75.4]

ADVERSE EVENTS:
Description: The same event may have appeared as both an adverse event (AE) and a serious AE (SAE). However, what was presented were distinct events. An event may have been categorized as serious in 1 subject and as nonserious in another subject, or 1 subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 13/83
Other Adverse Events (participants affected / at risk) | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=83)
Dehydration (Metabolism and nutrition disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Confusional state (Psychiatric disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Anal abscess (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Aphasia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=83)
Anaemia (Blood and lymphatic system disorders) | 20
Leukopenia (Blood and lymphatic system disorders) | 33
Neutropenia (Blood and lymphatic system disorders) | 37
Thrombocytopenia (Blood and lymphatic system disorders) | 34
Hypothyroidism (Endocrine disorders) | 8
Lacrimation increased (Eye disorders) | 5
Vision blurred (Eye disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 44
Dry mouth (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9
Glossodynia (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 40
Oral pain (Gastrointestinal disorders) | 12
Stomatitis (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 27
Asthenia (General disorders) | 9
Fatigue (General disorders) | 50
Mucosal inflammation (General disorders) | 5
Pyrexia (General disorders) | 5
Urinary tract infection (Infections and infestations) | 12
Contusion (Injury, poisoning and procedural complications) | 7
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 10
Blood alkaline phosphatase increased (Investigations) | 7
Blood creatinine increased (Investigations) | 5
Weight decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 36
Dehydration (Metabolism and nutrition disorders) | 13
Hypokalaemia (Metabolism and nutrition disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 26
Headache (Nervous system disorders) | 14
Insomnia (Psychiatric disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Acne (Skin and subcutaneous tissue disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 9
Hair colour changes (Skin and subcutaneous tissue disorders) | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 17
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 14
Skin discolouration (Skin and subcutaneous tissue disorders) | 5
Yellow skin (Skin and subcutaneous tissue disorders) | 11
Hypertension (Vascular disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.